CLINICAL TRIAL: NCT00152945
Title: Determining the Responsiveness of Intestinal Lipoprotein Production to an Elevation of Plasma Free Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Gary Lewis, Professor, Department of Medicine and Physiology, University Health Network, Toronto
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-0575-B; CIHR Grant 777509574
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Insulin Resistance
Keywords: intestinal lipoprotein; very low density lipoprotein; free fatty acids; Apo B48 and Apo B100; triglycerides; Intestinal lipoprotein production
MeSH Terms: conditions — Insulin Resistance | interventions — Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravenous Intralipid — intravenous infusion
Drug: Intravenous leucine, glycerol — intravenous infusion

SUMMARY:
Lipoproteins are large complexes of molecules that transport lipids (primarily triglycerides and cholesterol) through the blood. The intestine has traditionally been viewed as a 'passive' organ with respect to lipoprotein production, with intestinal lipoprotein production rates responding mainly to fat ingestion and absorption. The investigators have recently demonstrated in animal models that there is an overproduction of intestinal lipoproteins in both the fasted and the fed state. The investigators have also recently demonstrated that an elevation of plasma free fatty acids (FFAs) stimulates intestinal lipoprotein in hamsters. It is not known whether intestinal lipoprotein production can be acutely stimulated by an elevation of plasma FFAs in humans.

Hypothesis: Intestinal lipoprotein particle production in humans can be stimulated by an acute elevation of plasma free fatty acids.

DETAILED DESCRIPTION:
This study proposes to use a published stable isotope method to study the kinetics of apoB48 and apoB100 in the constant fed state in healthy subjects. These studies will be performed in 10 healthy, lean men and women aged 18 to 65 years of age. Each subject will serve as his/her own control and will undergo 3 separate lipoprotein turnover studies, in random order, 4 to 6 weeks apart. Since the infusion of intralipid (a synthetic triglyceride emulsion that provides a source of fatty acids) and heparin (to activate lipoprotein lipase) raises both FFAs and glycerol, two control studies will be performed, one with saline and one with glycerol infusion. ApoB48-containing lipoprotein particle production will be determined as outlined above but for this study in the fasted state, in response to the following interventions:

1. Intralipid (20% solution @ 40 ml/hr) and heparin (250 u/hr) infusion to achieve an ~2-fold elevation of plasma FFAs (as previously shown), starting 90 minutes prior to and continuing throughout the lipoprotein turnover experiment,
2. Saline infusion control study, and
3. Glycerol control study in which glycerol will be infused at a rate of 2.25 g/hr to simulate the infusion of glycerol contained in Intralipid.

Stable isotope infusion protocol. Following a 14-h overnight fast, an IV will be inserted into a superficial vein in each forearm, one for infusion and one for sampling. At 7 am, a fasting blood sample will be drawn and the subject will begin to ingest the first of 15 identical small hourly meals, each equivalent to 1/15th of their daily food intake. This will be achieved by giving the patient the drink BOOST (Mead Johnson Nutritionals, Ottawa, On) and, using the Harris Benedict Equation (HBE) to determine the number of total energy requirements. This is based on height, weight, age and activity factors. The subject will have nothing else to eat until the end of the study. At the same time an IV infusion with either heparin plus intralipid or saline or glycerol as indicated above will be started. At 10 am (3 hours after starting the ingestion of hourly feeds), a primed-constant infusion of deuterium-labeled leucine ([D3]L-leucine 98%, Cambridge Isotope Laboratories, MA) will be started, as previously described (0.6 mg/kg as an initial injection and then 0.6 mg/kg/hr thereafter). In addition, an IV bolus of d5-glycerol (100 mmol/kg) will be administered. These are standard techniques used for the assessment of lipoprotein metabolism in humans. Leucine, an amino acid and glycerol, an intermediary metabolite, are used by cells in the body as building blocks for proteins, fats and for energy. The form of leucine that will be administered is deuterated leucine (chemical formula L-[5,5,5-2H3]) and the form of glycerol is d5-glycerol, which has been enriched with the naturally occurring isotope (chemical variant) of hydrogen (2H). Deuterated leucine and glycerol are stable isotopes that occur naturally in the environment and in the body, and there are no health/safety issues regarding the infusion of the amounts of deuterated leucine and glycerol indicated above. The solutions are prepared using sterile techniques and are monitored for contamination prior to administration. Blood samples will be collected prior to and at the following time points after administration of the stable isotopes: 1hr, 2hr, 3hr, 5hr, 7hr, 9hr, 10hr, 11hr and 12hr. A total of 340 ml of blood will be drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Non-diabetic men and women aged 18-65 years old
2. Written informed consent obtained
3. Body mass index (BMI) < 27 kg/m2
4. Fasting triglycerides < 2.5 mmol/l
5. Waist circumference < 90 cm
6. Fasting blood glucose < 6 mmol/l
7. Haemoglobin above 130 g/L.

Exclusion Criteria:

1. Patient has a history of hepatitis/hepatic disease that has been active within the previous 2 years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (creatinine [Cr] > 1.5 mg/dL) genitourinary, or hematological systems; or severe uncontrolled treated or untreated hypertension (sitting diastolic blood pressure [BP] > 100 or systolic > 180); or proliferative retinopathy.
3. Fasting blood glucose > 6 mmol/l or known diabetes.
4. Any history of a myocardial infarction (MI) or clinically significant, active, cardiovascular history including a history of arrhythmias or conduction delays on electrocardiogram (ECG), unstable angina, or decompensated heart failure.
5. Any laboratory values: AST > 2x upper limit of normal (ULN); ALT > 2x ULN; thyroid-stimulating hormone (TSH) > 6 mU/l.
6. Known or suspected allergy to the medication or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions.
7. Current addiction to alcohol or substances of abuse as determined by the investigator.
8. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
9. Any lipid lowering or hypoglycemic agents
10. Will not donate blood three months before start or three months after completing study.
11. Thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine if the elevation of plasma FFAs by infusing intralipid and heparin stimulates intestinal lipoprotein production | blood samples at 1,2,3,5,7,9,10,11 and 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Lewis, MD, Principal Investigator — University Health Network, Toronto, Ontario, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada